CLINICAL TRIAL: NCT04168970
Title: Percutaneous Left Stellate Ganglion Block In Out-of-hospital Cardiac Arrest Due to Refractory VEntricular Arrhythmias
Brief Title: Percutaneous Left Stellate Ganglion Block In Out-of-hospital Cardiac Arrest Due to Refractory VEntricular Arrhythmias (LIVE Study)
Acronym: LIVE
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Azienda Regionale Emergenza Urgenza (AREU) (Unknown); University of Pavia (Other)
Responsible Party: Principal Investigator, Simone Savastano, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: LIVE Study
Record Dates: First submitted 2019-09-14; First posted 2019-11-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Ventricular Fibrillation Sustained
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSGB group: MD will perform PSGB using Lidocaine. The PGSB will be performed after the administration of the 4th shock if the 3rd shock was unsuccessful in restoring a stable perfusing rhythm, considering all the shocks administered both by an AED or by manual defibrillator. PSGB will be performed after all the actions provided in the ACLS algorithm and which are considered useful in the clinical situation (intubation and ventilation, administration of iv/io adrenaline, amiodarone or lidocaine, use of mechanical chest compression, etc.).
  Interventions: Procedure: PSGB
- Control group: Historical cohort of patients with the same OHCA characteristics (first shockable rhythm and who received more than 4 shocks) enrolled in the Cardiac Arrest Registry of the Province of Pavia

INTERVENTIONS:
Procedure: PSGB — Percutaneous stellate ganglion block: injection of 10 mL of local anaesthetic (lidocaine 2%) at the C6 level using the anatomic technique or the echo-guided technique The anaesthetic that will be used for PSGB is lidocaine.
  Groups: PSGB group

SUMMARY:
A prospective uncontrolled study to verify the feasibility and practicability of percutaneous stellate ganglion block (PSGB) in patient suffering from a refractory out-of-hospital cardiac arrest (OHCA) due to a shockable rhythm and the eventual occurrence of complication related to it. The study will also assess whether the rate of return of spontaneous circulation (ROSC) until admission and transfer of care to the receiving hospital is higher in the patients treated with PSGB as compared to historical controls.

DETAILED DESCRIPTION:
This is a prospective uncontrolled study. All patients meeting the inclusion criteria will be consecutively enrolled in the study. The Emergency Medical System (EMS) rescue team medical doctor (MD) will be asked to perform PSGB after all the actions provided in the ACLS algorithm and which are considered useful in the clinical situation (intubation and ventilation, administration of iv/io adrenaline, amiodarone or lidocaine, use of mechanical chest compression, etc.). The PGSB will be performed after the administration of the 4th shock if the 3rd shock was unsuccessful in restoring a stable perfusing rhythm, considering all the shocks administered both by an AED or by manual defibrillator. The evaluation of the effectiveness of the 3rd shock will be carried out at the end of the two-minute cycle after shock delivery, as recommended by the guidelines. If the MD will arrive on the scene after the delivery of the 3rd shock, the PSGB should be executed as soon as possible after performing all the actions which are considered useful in the clinical situation. The MD, based on his confidence, can choose to use the anatomic technique or the echo-guided technique. The technique will be performed in the pre-hospital setting. Those patients with refractory OHCA transported with ongoing ACLS who receive the fourth shock once in the emergency department will be also considered. On the contrary patients with prehospital ROSC who suffer a new cardiac arrest once in the emergency department won't be considered in the present study. The MD will be asked to evaluate the presence of anisocoria immediately before the PSGB and 1-2 minutes after the PSGB. In case of absence of anisocoria 2 minutes after PSGB, MD can try PSGB another time. The anaesthetic that will be used for PSGB is lidocaine 2%, which is already available among EMS drugs. After the end of the event, the MD will be asked to fill in a questionnaire regarding the feasibility of the technique in the pre-hospital setting, the practicability of its implementation compared to the usual procedures performed in the pre-hospital setting and any problems encountered. The responses will be scored from 1 to 10 (1=perfect feasibility; 10=no feasibility). All eventual complications associated with PSGB will be carefully recorded.

The effectiveness of the PSGB will be evaluated if at least one shock will be delivered after the execution of PSGB.

The data will be compared to our historical cohort of patients with the same OHCA characteristics (first shockable rhythm and who received more than 4 shocks) enrolled in the Cardiac Arrest Registry of the Province of Pavia from 1 January 2016 to 31 December 2017.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an OHCA occurred in the Province of Pavia in which the first rhythm was a shockable one

Exclusion Criteria:

* Patients in which the cause of the cardiac arrest is non-medical following Utstein-style 2014 (trauma, overdose, drowning, electrocution, asphyxia)
* Patients who has an anisocoria at the arrival of medical doctor on the scene
* Patients whose neck is judge unsuitable for PSGB by the operator (i.e. presence of big scar, thyroid goiter, etc.)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an OHCA occurred in the Province of Pavia in which the first rhythm was a shockable one and with at least three episode of VT/VF during the out-of-hospital resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | Up to hospital discharge (on average 15 days after the event)
  The occurrence of complications associated with PSGB in the pre-hospital setting
Feasibility of PSGB in the pre-hospital setting | Up to 24 hours after the event
  The feasibility and practicability of PSGB in the pre-hospital setting based on a questionnaire filled out by the physician who performed the PSGB
Survived event | Up to hospital admission
  To assess whether the rate of ROSC until admission and transfer of care to the receiving hospital is higher in the patients treated with PSGB as compared to historical controls.

SECONDARY OUTCOMES:
Rate of rhythm conversion after first defibrillation | During resuscitation
  The rate of rhythm conversion at the first defibrillation after the PSGB
Rate of rhythm conversion after second defibrillation | During resuscitation
  The rate of rhythm conversion at the second defibrillation after the PSGB
Rate of ROSC if anisocoria is present | Up to hospital admission
  To assess whether the rate of ROSC is higher in the patients treated with PSGB and in which anisocoria is present after the PSGB, but not before PSGB
Rate of ROSC | Up to hospital admission
  To assess whether the rate of ROSC is higher in the patients treated with PSGB
Survived event if anisocoria present | Up to hospital admission
  To assess whether the rate of ROSC until admission and transfer of care to the receiving hospital is higher in the patients treated with PSGB and in which anisocoria is present after the PSGB, but not before PSGB
Survival at hospital discharge | Up to hospital discharge (on average 15 days after the event)
  To assess whether the survival rate at hospital discharge is higher in the patients treated with PSGB.
Survival at hospital discharge if anisocoria present | Up to hospital discharge (on average 15 days after the event)
  To assess whether the survival rate at hospital discharge is higher in the patients treated with PSGB and in which anisocoria is present after the PSGB, but not before PSGB
Survival with good neurological outcome | 1 month after the cardiac arrest
  To assess whether the survival rate with good neurological outcome (CPC 1 ore 2) at 1 month after the event is higher in the patients treated with PSGB
Survival with good neurological outcome if anisocoria present | 1 month after the cardiac arrest
  To assess whether the survival rate with good neurological outcome (CPC 1 ore 2) at 1 month after the event is higher in the patients treated with PSGB and in which anisocoria is present after the PSGB, but not before PSGB.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT04168970/Prot_SAP_000.pdf